CLINICAL TRIAL: NCT00816738
Title: Evaluation of the Treatment of Recurrent Corneal Erosions by Anterior Stromal Puncture With Nd: YAG Laser
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yu-Chih Hou/Department of Ophthalmology, National Taiwan University Hospital, Organization: Department of Ophthalmology, National Taiwan University Hospital
Other Study IDs: 200801035R
Record Dates: First submitted 2008-08-31; First posted 2009-01-05 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: Recurrent Corneal Erosion; Trauma
Keywords: Nd: YAG laser; recurrent corneal erosions; trauma; anterior stromal puncture
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the clinical outcomes in patients with recurrent corneal erosions who received anterior stromal puncture by use of neodymium:yttrium-aluminum-garnet (Nd:YAG) laser.

DETAILED DESCRIPTION:
Participants: From 2000 to 2005, thirty-three eyes in 33 patients with unilaterally recurrent corneal erosions who showed poor response to conservative managements and were treated with Nd:YAG laser were studied.

Intervention: Anterior corneal stromal puncture with Nd:YAG laser was performed in the loosened epithelium or epithelial defect area. The causes and frequency of corneal erosions and the spot numbers and total energy of the Nd:YAG laser were recorded. Slit-lamp biomicroscopic examination, refraction, corneal topography, and times of laser were reviewed. A questionnaire regarding the preoperative and postoperative difference in the intensity of pain and frequency of corneal erosion was provided.

Main Outcome Measures: Rate of recurrence and pain assessment by numerical rating scale.

ELIGIBILITY:
Inclusion Criteria:

* patients with recurrent corneal erosions who showed poor response to conservative managements and were treated with Nd:YAG laser.

Exclusion Criteria:

* Slit-lamp biomicroscopic examination in both eyes of patient showed any evidence of anterior basement membrane dystrophy.

Ages: 20 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: to evaluate the clinical outcomes after anterior stromal puncture with Nd:YAG laser in a consecutive series of 33 eyes in 33 patients with unilaterally recurrent corneal erosion.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2008-01; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Cure rate of recurrent corneal erosions (frequency of attack and numbers of Nd: YAG laser treatment), intensity of pain relief and visual acuity. | Before treatment, weekly after the treatment, and monthly after symptom relief

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chih Ho, MD, Study Director — National Taiwan University Hospital; Tzu-Hsun Tsai, MD, Principal Investigator — National Taiwan University Hospital; Tzu-Yun Tsai, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan